CLINICAL TRIAL: NCT06343714
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of Escalating Single and Multiple Doses of FB1003 in the Healthy and Osteoarthritis Pain Subjects
Brief Title: A Study of FB1003 in Healthy and Osteoarthritis Pain Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: 4B Technologies Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FB1003-04-101
Record Dates: First submitted 2024-03-14; First posted 2024-04-03 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteers
Keywords: Healthy participants, Osteoarthritis pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- SAD Cohort 1 (Experimental): Participants in this cohort will receive SAD dose 1 of FB1003 or Placebo.
  Interventions: Drug: FB1003; Drug: Placebo
- SAD Cohort 2 (Experimental): Participants in this cohort will receive SAD dose 2 of FB1003 or Placebo.
  Interventions: Drug: FB1003; Drug: Placebo
- SAD Cohort 3 (Experimental): Participants in this cohort will receive SAD dose 3 of FB1003 or Placebo.
  Interventions: Drug: FB1003; Drug: Placebo
- SAD Cohort 4 (Experimental): Participants in this cohort will receive SAD dose 4 of FB1003 or Placebo.
  Interventions: Drug: FB1003; Drug: Placebo
- SAD Cohort 5 (Experimental): Participants in this cohort will receive SAD dose 5 of FB1003 or Placebo.
  Interventions: Drug: FB1003; Drug: Placebo
- OA pain Cohort1 (Experimental): Participants in this cohort will receive OA pain dose 1 of FB1003 or Placebo.
  Interventions: Drug: FB1003; Drug: Placebo
- OA pain Cohort 2 (Experimental): Participants in this cohort will receive OA pain dose 2 of FB1003 or Placebo.
  Interventions: Drug: FB1003; Drug: Placebo
- OA pain Cohort 3 (Experimental): Participants in this cohort will receive OA pain dose 3 of FB1003 or Placebo.
  Interventions: Drug: FB1003; Drug: Placebo

INTERVENTIONS:
Drug: FB1003 — Subcutaneous (SC) injection
Drug: Placebo — Subcutaneous (SC) injection

SUMMARY:
The purpose of Part 1 is to evaluate safety and tolerability of FB1003 when given subcutaneously to healthy participants. Blood tests will be done to examine blood exposure, concentration and half-life of FB1003 following administrations. For each participant, the study will last up to about 12 weeks for single ascending dose part, and 18 weeks for multiple ascending dose part, including screening.

The purpose of Part 2 is to assess the safety, tolerability, PK and efficacy of SAD of SC administered FB1003 in adult subjects with osteoarthritis (OA) pain.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects who, at the time of signing the informed consent form (ICF), are between 18 and 55 years of age (inclusive).
* The subject is capable of understanding and complying with protocol requirements
* Subjects in good health based on pre-study medical history, physical examinations, vital signs, abdominal ultrasound, 12-lead ECGs, clinical laboratory tests.
* Be willing to refrain from taking NSAID medications for 1 week prior to receiving study intervention and for 2 weeks after study intervention administration.
* The subject weighs at least 45 kg and has a body mass index between 18 and 32 kg/m2 (inclusive).
* Must be capable of giving signed informed consent as described which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
* Women not of childbearing potential. OR must agree to use a double barrier highly effective method of contraception from the beginning of screening until at least 90 days after the last dose of study intervention.

DISEASE CONDITIONS (PART 2 ONLY)

* Subject has confirmation of OA of the knee through the radiographs of both knees with a Posterior-Anterior, Fixed-flexion view taken during the Screening Period using American College of Rheumatology (ACR) clinical and radiographic diagnostic criteria.
* Evidence of knee OA with a Kellgren and Lawrence (KL) Grade ≥2.
* Subject is willing to discontinue all pain medication at least 5 half-lives from Day 1 visit and agree to take only the allowed Rescue Medications through study completion (maximum 4000 mg paracetamol per day).
* Subject has moderate to severe pain in the index joint defined as a Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) average pain subscale score of ≥4 at both the screening and randomization visits.

Exclusion Criteria:

* Medical conditions for Part 1 only:

  1. History or presence at the screening visit of bone or joint disorders including but not limited to OA, avascular necrosis, destructive arthropathy, pathologic fractures, osteonecrosis, rheumatoid arthritis, neuropathic joint arthropathy, lupus erythematosus, or inflammatory joint diseases.
  2. History of joint-related events such as, but not limited to, total joint replacement surgery, patella dislocation, hip dislocation, knee dislocation, or joint infections.
  3. Trauma to any joint in the 30 days prior to the screening visit.
* Medical conditions for Part 2 only:

  1. Clinically significant hematological findings at screening.
  2. Abnormal findings indicating renal impairment, such as creatinine ≥1.5×ULN, estimated glomerular filtration rate (eGFR) of ≤60 mL/min/1.73 m2 in adults, as calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula, at screening.
  3. A history of non-febrile seizures.
  4. History of inflammatory arthritis other than OA, in the judgment of the investigator would make the subject inappropriate for entry into this study.
  5. History of osteonecrosis / osteoporotic fracture (including minimally traumatic or atraumatic fracture).
  6. History of significant trauma (including sports injury) or surgery to a knee, hip or shoulder within last year.
  7. Fibromyalgia, regional pain caused by lumbar / cervical compression with radiculopathy, or other moderate/severe pain that may confound assessment of knee pain.
  8. A hospital admission or major surgery within 60 days prior to screening.
  9. Planned surgery to a knee, hip, or shoulder during the study.
* Active or history of serious mental illness or psychiatric disorder, including but not limited to schizophrenia, bipolar disorder, or major depressive disorder, which require current medical intervention.
* Subject has abnormal screening or Check-in (D-1) laboratory values that suggest a clinically significant underlying disease or subject has the following lab abnormalities: alanine transferase (ALT) and/or aspartate transaminase (AST) >1.5 upper limit of normal (ULN).
* History of autonomic neuropathy, or diabetic neuropathy, or evidence of autonomic neuropathy, or presence of clinically relevant peripheral neuropathy.
* Resting heart rate of <50 or >100 beats per minute (not on ECG).
* History or evidence at screening of heart block.
* History of myocardial infarction, acute coronary syndromes, or cerebrovascular accident within 12 months prior to the screening visit.
* Human immunodeficiency virus (HIV), hepatitis B, or hepatitis C positive by serological testing at the screening visit.
* History or presence of malignancy within 5 years prior to screening, except subjects who have been treated successfully with no recurrence of basal or squamous cell carcinoma of the skin (<1 year), in situ cervical cancer, or in situ ductal breast cancer.
* Women of reproductive potential who have a positive serum pregnancy test result at the screening visit, or a positive urine pregnancy test result at the baseline visit (D-1), or who do not have their pregnancy test results on D-1.
* Subject has donated or lost 400 mL or more of his or her blood volume (including plasmapheresis) or had a transfusion of any blood product within 30 days prior to first dose of study intervention.
* Clinically significant illness within seven days before the first dose of the study intervention.
* History of multiple drug allergies or history of allergic reaction to the monoclonal antibody.
* History of severe intolerance to SC injection (minor reactions are permitted, e.g., localized swelling or redness).
* Significant concomitant illness or any medical or surgical condition, such as, but not limited to, cardiac, renal, neurological, endocrinological, gastrointestinal, hepatic, metabolic or lymphatic disease that would adversely affect the subject's participation in this study or interpretation of safety/PK data.
* Dosing with another investigational drug or therapy within 30 days or at least 5 half-lives of the investigational drug, whichever is longer.
* Systolic blood pressure (SBP) >140 mmHg and/or diastolic blood pressure (DBP) >90 mmHg after 5 minutes of resting in a seated position, unless determined by the Investigator to be not clinically relevant and well controlled with medications.
* Pregnant or breast-feeding women.
* Any conditions which would make the subject unsuitable for enrollment or could interfere with the subject's participation in or completion of the study in the opinion of the Investigator.
* Consume more than 14 (female) or 21 (male) units of alcohol per week (unit: 1 glass of wine (125 mL) = 1 measure of spirits = ½ pint of beer) within the 12 months before screening or positive screen for alcohol abuse.
* Smoking >4 cigarettes (or an equivalent amount of any other nicotine-containing product) per day within 30 days before screening.
* History or clinical evidence of drug abuse within the 12 months before screening or positive screen for drug abuse. Drug abuse is defined as compulsive, repetitive, and/or chronic use of drugs or other substances with or without problems related to their use and/or when stopping or a dose reduction will lead to withdrawal symptoms.
* Have received a live and/or non-live vaccine (including COVID) within 28 days prior to dosing or intend to receive a vaccine during the study period or at least 56 days after the last dose of IP.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-04-07 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint in the study is the incidence and severity of treatment emergent adverse events (TEAEs) in participants treated with FB1003 or placebo. | Baseline to end of study, SAD up to 56 days and MAD up to 84 days.
  The percentages of subjects experiencing AEs will be calculated.

SECONDARY OUTCOMES:
FB1003 serum concentrations over time | Baseline to end of study, SAD up to 56 days and MAD up to 84 days.
  The concentration of FB1003 will be evaluated.
PK: Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC0-∞) of FB1003 | Baseline to end of study, SAD up to 56 days and MAD up to 84 days.
  AUC0-∞ of FB1003 will be evaluated. The unit of measure is hour*microgram per milliliter (hr*mcg/mL).
Presence of anti-FB1003 antibodies over time | Baseline to end of study, SAD up to 56 days and MAD up to 84 days)
  The percentage of subjects testing positive for ADA will be calculated.
To assess the effect of FB1003 on overall changes of disease activity following SC administration in subjects with OA pain (Part 2). | 12 weeks.
  Efficacy endpoints include:
  * Changes from baseline in WOMAC pain, function and stiffness sub-scales during treatment
  * Changes from baseline in NRS scale during treatment

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Nucleus Network, Brisbane, Queensland
  - Veritus Research, Bayswater, Victoria

IPD SHARING:
Plan to Share IPD: No